CLINICAL TRIAL: NCT03454841
Title: Comparison of Circadian Variability of Platelet Inhibition in Patients With Myocardial Infarction Treated With Prasugrel and Ticagrelor
Brief Title: Daily Variability of Platelet Aggregation in Patients With Myocardial Infarction Treated With Prasugrel and Ticagrelor
Acronym: DRAGON
Status: Completed | Type: Observational
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Jacek Kubica, Prof. dr hab., Collegium Medicum w Bydgoszczy
Other Study IDs: CMUMK202I
Record Dates: First submitted 2018-02-27; First posted 2018-03-06 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Acute Myocardial Infarction
Keywords: prasugrel; ticagrelor; VASP; platelet reactivity; STEMI; NSTEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prasugrel: Patients with myocardial infarction will receive prasugrel as a part of dual antiplatelet therapy with aspirin.
  Interventions: Drug: Prasugrel
- Ticagrelor: Patients with myocardial infarction will receive ticagrelor as a part of dual antiplatelet therapy with aspirin.
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Prasugrel — Patients with myocardial infarction will receive a 60 mg prasugrel loading dose, followed by a maintenance dose of 10 mg once daily
  Other Names: Efient
  Groups: Prasugrel
Drug: Ticagrelor — Patients with myocardial infarction will receive a 180 mg ticagrelor loading dose, followed by a maintenance dose of 90 mg twice daily
  Other Names: Brilique
  Groups: Ticagrelor

SUMMARY:
The aim of this study is to compare circadian variability of antiplatelet effect of prasugrel and ticagrelor maintenance doses during the initial days after acute myocardial infarction.

DETAILED DESCRIPTION:
Prasugrel and ticagrelor are two oral P2Y12 receptor antagonists recommended as a part of dual antiplatelet therapy with aspirin in patients with acute myocardial infarction. Both drugs exert comparable antiplatelet effect following a loading dose. However, pharmacodynamic differences exist between these P2Y12 receptor inhibitors. Prasugrel is a prodrug that requires hepatic activation and permanently binds to platelet P2Y12 receptors, whereas ticagrelor is an active drug and blocks P2Y12 receptors reversibly. Another important difference is that prasugrel maintenance dose is administered once daily, while ticagrelor requires next dosage every 12 hours. These fundamental distinctions may affect the degree of platelet inhibition on maintenance doses during the first days after acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* provision of informed consent prior to any study specific procedures
* diagnosis of acute ST-segment elevation myocardial infarction or acute non-ST-segment elevation myocardial infarction
* male or non-pregnant female, aged 18-75 years old
* provision of informed consent for angiography and percutaneous coronary intervention

Exclusion Criteria:

* treatment with ticlopidine, clopidogrel, prasugrel or ticagrelor within 14 days before the study enrollment
* hypersensitivity to ticagrelor or prasugrel
* contraindications for ticagrelor or prasugrel
* current treatment with oral anticoagulant or chronic therapy with low-molecular-weight heparin
* active bleeding
* history of ischemic stroke or transient ischemic attack
* history of intracranial hemorrhage
* recent gastrointestinal bleeding (within 30 days)
* history of moderate or severe hepatic impairment
* history of major surgery or severe trauma (within 3 months)
* patient required dialysis
* manifest infection or inflammatory state
* concomitant therapy with strong CYP3A inhibitors (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir) or strong CYP3A inducers (rifampicin, phenytoin, carbamazepine, dexamethasone, phenobarbital) within 14 days and during study treatment
* body weight below 60 kg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute myocardial infarction treated invasively.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Circadian variability of platelet inhibition assessed with VASP | Day 4 after acute myocardial infarction
  Platelet inhibition evaluated with VASP assay at 8:00, 12:00, 16:00 and 20:00
Circadian variability of platelet inhibition assessed with Multiplate | Day 4 after acute myocardial infarction
  Platelet inhibition evaluated with Multiplate at 8:00, 12:00, 16:00 and 20:00

SECONDARY OUTCOMES:
High platelet reactivity at 8:00 assessed with VASP | Day 4 after acute myocardial infarction
  Number of patients with high platelet reactivity evaluated with VASP assay at 8:00
High platelet reactivity at 12:00 assessed with VASP | Day 4 after acute myocardial infarction
  Number of patients with high platelet reactivity evaluated with VASP assay at 12:00
High platelet reactivity 16:00 assessed with VASP | Day 4 after acute myocardial infarction
  Number of patients with high platelet reactivity evaluated with VASP assay at 16:00
High platelet reactivity 20:00 assessed with VASP | Day 4 after acute myocardial infarction
  Number of patients with high platelet reactivity evaluated with VASP assay at 20:00
High platelet reactivity 08:00 assessed with Multiplate | Day 4 after acute myocardial infarction
  Number of patients with high platelet reactivity evaluated with Multiplate at 08:00
High platelet reactivity 12:00 assessed with Multiplate | Day 4 after acute myocardial infarction
  Number of patients with high platelet reactivity evaluated with Multiplate at 12:00
High platelet reactivity 16:00 assessed with Multiplate | Day 4 after acute myocardial infarction
  Number of patients with high platelet reactivity evaluated with Multiplate at 16:00
High platelet reactivity 20:00 assessed with Multiplate | Day 4 after acute myocardial infarction
  Number of patients with high platelet reactivity evaluated with Multiplate at 20:00

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Kubica, Prof., Principal Investigator — Department of Cardiology and Internal Medicine, Collegium Medicum, Nicolaus Copernicus University, Bydgoszcz, Poland
Locations (2):
- Poland (2):
  - Department of Cardiology, Dr. A. Jurasz University Hospital, Collegium Medicum, Nicolaus Copernicus University, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Department of Cardiology, Wrocław Medical University, Wroclaw, Lower Silesian Voivodeship